CLINICAL TRIAL: NCT03350126
Title: Interest of iRECIST Radiological Assessment for Disease Control Rate (DCR) for Evaluation of Patients With Metastatic Colorectal Cancer dMMR and/or MSI Treated With Nivolumab and Ipilimumab. A GERCOR Open-label Phase II Study NIPICOL C17-01
Brief Title: iRECIST Evaluation's Relevance for DCR in MMR/MSI Metastatic Colorectal Cancer Patients on Nivolumab and Ipilimumab
Acronym: NIPICOL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIPICOL C17-01
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Cancer Colorectal
Keywords: MSI or MMR
MeSH Terms: conditions — Colonic Neoplasms; Microsatellite Instability | interventions — Ipilimumab; Injections; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Therapy induction (12 weeks) Nivolumab (IV) and Ipilimumab (IV) - every 21 days - 4 cycles Then Nivolumab (IV) alone every 15 days - 20 cycles - until 12 months
  Interventions: Drug: Ipilimumab 200 MG in 40 ML Injection; Drug: Nivolumab 10 MG/ML

INTERVENTIONS:
Drug: Ipilimumab 200 MG in 40 ML Injection — Induction therapy (12 weeks):
  Nivolumab 3mg/kg intravenously (IV) over 60 minutes and Ipilimumab 1mg/kg (IV) over 90 minutes Q3W
Drug: Nivolumab 10 MG/ML — Induction therapy (12 weeks) :
  Nivolumab 3mg/kg intravenously (IV) over 60 minutes and Ipilimumab 1mg/kg (IV) over 90 minutes Q3W
  Maintenance therapy (40 weeks):
  Nivolumab monotherapy IV over 60 minutes Q2W until iRECIST progression or if no PD for one year.

SUMMARY:
This is a non-randomized study, open label phase II study. The purpose of this study is to evaluate disease control rate (DCR) by RECIST and iRECIST at 12 weeks.

Evaluation of RECIST and iRECIST will be done in each center in order to choose the optimal therapy (Assessment by Investigators).

A centralized evaluation of RECIST and iRECIST, will be organized in Saint-Antoine.

DETAILED DESCRIPTION:
Recent studies have shown sensitivity to immunotherapy treatment in patients with metastatic colorectal cancer with a dMMR tumor. The association nivolumab plus ipilimumab demonstrated encouraging results with durable responses in these patients.

The criteria for assessing responses for solid tumors are currently based on RECIST 1.1, which are well correlated with the clinical response to chemotherapy. However, in patients treated with immunotherapy, such criteria are less accurate, as already demonstrated in the treatment of metastatic melanoma, but not yet in other malignant tumors.

Therefore, we hope with this study, to identify more accurate imaging criteria that could help oncologists to make optimal decisions for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study drug,
3. Men and women are required to use adequate birth control during the study (when applicable):

   Within the frame of this study, female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control (i.e., pregnancy rate of less than 1% per year) during the period of treatment and for 5 months for women and 7 months for men from the last treatment administration. Men must refrain from donating sperm during this same period.

   Contraceptive methods that result in a low failure rate when used consistently and correctly include methods such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intrauterine devices, intrauterine hormone-releasing stem, true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant), bilateral tubal occlusion, or a female partner who is not of childbearing potential or a male partner who has had a vasectomy. Women and female partners using hormonal contraceptive must also use a barrier method i.e. condom or occlusive cap (diaphragm or cervical/vault caps).

   A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
4. Histologically proven metastatic adenocarcinoma of the colon and/or rectum,
5. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study,
6. dMMR DNA (protein expression by ICH and/or MSI by PCR):

   * Tumor MMR and/or MSI will be assessed per local guidelines: ICH with two (anti-MLH1 and anti-MSH2) or four antibodies (anti-MLH1, anti-MSH2, anti-MSH6 and anti-PMS2) and/or PCR (with PROMEGA: BAT25, BAT26, NR21, NR24, NR27]) by the investigators prior to screening,
   * In ICH, the extinction of MLH1 (+/- PMS2), or MSH2 (+/- MSH6), or MSH6, or PMS2 alone is necessary for inclusion (dMMR),
   * In PCR, we recommended pentaplex panel (BAT25, BAT26, NR21, NR24, and NR27). Tumor samples with instability in 0, 1, or ≥2 markers were identified as MSS, MSI-L, and MSI-H, respectively. Only tumor samples with ≥2 instable markers are necessary for inclusion (MSI-H).

   Agreement of the SPONSOR (GERCOR) will be mandatory to include a patient. GERCOR will check every patient's file to confirm the dMMR/ MSI-H patient's status before inclusion (an anonymized fax. The confirmation of a patient's allocation will be immediately sent by mail to the investigator).
7. Age ≥18 years,
8. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1,
9. Progression during, after, or who are intolerant or have contraindication to approved standard therapies for the metastatic disease which must include at least:

   * Fluoropyrimidine, and oxaliplatin and irinotecan.
   * Anti-EGFR therapy if wild-type RAS and RAF and anti-VEGF therapy,
10. Hematological status: absolute neutrophil count (ANC) ≥1.5x109/L; platelets ≥100x109/L; hemoglobin ≥9g/dL,
11. Adequate renal function: serum creatinine level <150µM,
12. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase <5xULN, alanine aminotransferase (ALAT) and aspartame aminotransferase (ASAT) ≤3.0x ULN (≤5.0x ULN for patients with liver involvement of their cancer),
13. Registration in a National Health Care System (CMU included),
14. Subjects must have measurable disease per RECIST 1.1. Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately,
15. Subject willing to comply to provide primary and metastatic tumor tissue (archival or fresh biopsy specimen), including possible pre-treatment biopsy, for PD-L1 expression analysis and other biomarker correlative studies,
16. At least one target lesion on CT,
17. No contraindication to Iodine contrast media injection during CT

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
2. Unresolved toxicity higher than Grade 1, NCI-CTCAE v 4.03, attributed to any prior therapy
3. Treatment with any investigational medicinal product within 28 days prior to study entry,
4. Major surgical procedure within 4 weeks prior to initiation of study treatment,
5. Other serious and uncontrolled non-malignant disease (including active infection),
6. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
7. Pregnant or breastfeeding women,
8. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.

   Note: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
9. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest imaging,
10. Human immunodeficiency virus (HIV),
11. Active hepatitis B virus (HBV, defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C virus (HCV), Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.

    Note: Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
12. Administration of a live, attenuated vaccine within four weeks prior to start of treatment or anticipation that such a live attenuated vaccine will be required during the remainder of the study,
13. Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents,
14. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within four weeks or five half-lives of the drug, whichever is shorter, prior to start of maintenance treatment,
15. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
16. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to start of maintenance treatment, or requirement for systemic immunosuppressive medications during the remainder of the study. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the Medical Monitor.

Note: Subjects are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Adrenal replacement steroid doses including doses >10 mg daily prednisone are permitted. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | At 12 weeks
  According with RECIST 1.1 and iRECIST

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | PFS is defined as time from date of first dose of study treatment to date of first Progression (accordance with RECIST 1.1 or iRECIST) or death due to any cause - Up to 24 months
  According with RECIST and iRECIST
Overall Response Rate (ORR) | Up to 24 months
  According with RECIST and iRECIST
Overall Survival (OS) | Up to 24 months
  OS is defined as the time between the date of the first dose of study treatment and the death date
Toxicity according to NCI-CTCAE version 4.0 (National Cancer Institute Common Terminology Criteria for Adverse Events), | Up to 24 months
  Patients will be assessed for AEs every visits and evaluations, PD, and treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, MD, Principal Investigator — Hopital Saint Antoine
Locations (8):
- France (8):
  - Institut Sainte Catherine, Avignon
  - CHRU Besançon, Besançon
  - Henri Mondor Hospital, Créteil
  - IHFB, Levallois-Perret
  - Centre Leon Berard, Lyon
  - CHU Nantes - Hôtel Dieu, Nantes
  - Hospital Saint Antoine, Paris
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Depotte L, Nay P, Borg C, Meurisse A, Henriques J, Bennouna J, De La Fouchardiere C, Tougeron D, Mazard T, Chibaudel B, Tournigand C, Vernerey D, Pigneur F, Andre T, Cohen R. Interplay between sarcopenia, GDF-15, and the efficacy of nivolumab plus ipilimumab in patients with mismatch repair deficient metastatic colorectal cancer: final survival analysis of the phase II GERCOR NIPICOL study. J Immunother Cancer. 2025 May 19;13(5):e011220. doi: 10.1136/jitc-2024-011220. PMID 40389373
- [Derived] Ratovomanana T, Nicolle R, Cohen R, Diehl A, Siret A, Letourneur Q, Buhard O, Perrier A, Guillerm E, Coulet F, Cervera P, Benusiglio P, Labreche K, Colle R, Collura A, Despras E, Le Rouzic P, Renaud F, Cros J, Alentorn A, Touat M, Ayadi M, Bourgoin P, Prunier C, Tournigand C, Fouchardiere C, Tougeron D, Jonchere V, Bennouna J, de Reynies A, Flejou JF, Svrcek M, Andre T, Duval A. Prediction of response to immune checkpoint blockade in patients with metastatic colorectal cancer with microsatellite instability. Ann Oncol. 2023 Aug;34(8):703-713. doi: 10.1016/j.annonc.2023.05.010. Epub 2023 Jun 1. PMID 37269904
- [Derived] Ratovomanana T, Cohen R, Svrcek M, Renaud F, Cervera P, Siret A, Letourneur Q, Buhard O, Bourgoin P, Guillerm E, Dorard C, Nicolle R, Ayadi M, Touat M, Bielle F, Sanson M, Le Rouzic P, Buisine MP, Piessen G, Collura A, Flejou JF, de Reynies A, Coulet F, Ghiringhelli F, Andre T, Jonchere V, Duval A. Performance of Next-Generation Sequencing for the Detection of Microsatellite Instability in Colorectal Cancer With Deficient DNA Mismatch Repair. Gastroenterology. 2021 Sep;161(3):814-826.e7. doi: 10.1053/j.gastro.2021.05.007. Epub 2021 May 13. PMID 33992635
- [Derived] Cohen R, Bennouna J, Meurisse A, Tournigand C, De La Fouchardiere C, Tougeron D, Borg C, Mazard T, Chibaudel B, Garcia-Larnicol ML, Svrcek M, Vernerey D, Menu Y, Andre T. RECIST and iRECIST criteria for the evaluation of nivolumab plus ipilimumab in patients with microsatellite instability-high/mismatch repair-deficient metastatic colorectal cancer: the GERCOR NIPICOL phase II study. J Immunother Cancer. 2020 Nov;8(2):e001499. doi: 10.1136/jitc-2020-001499. PMID 33148693